CLINICAL TRIAL: NCT01771601
Title: Cerebral Oximetry in Newborns - Comparing INVOS 5100c and OxyPrem vs. 1.2's Absolute Values, Sensitivity for Low Oxygen Levels and Reproducibility
Brief Title: Cerebral Oximetry in Newborns - Comparing INVOS 5100c and OxyPrem vs. 1.2
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other)
Responsible Party: Principal Investigator, Gorm Greisen, professor, Rigshospitalet, Denmark
Other Study IDs: 090113OXYVOS
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Near-infrared Spectroscopy, Transition, Caesarean Section
Keywords: Near-infrared spectroscopy, cerebral oxygenation, term newborn, reproducibility,

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Near-infrared spectroscopy sensors: Term infants born by elective Caesarean section

SUMMARY:
Regional tissue oxygenation (cStO2) can be monitored by near infrared spectroscopy. The commercial device INVOS 5100 (COVIDIEN, Mansfield, MA, USA) and the prototype OxyPrem vs. 1.2 (Biomedical Optics Research Laboratory, Zurich, Switzerland) will be used simultaneously to test for their relative sensitivity for low oxygen levels just after birth on term infants born by elective caesarean section. Reproducibility will be examined by replacements of the sensors six times the next day when the infant is stable and quiet. The Adult Somasensor (INVOS) will be used together with the OxyPrem sensor.

ELIGIBILITY:
Inclusion Criteria:

* Term infants
* Elective caesarean section

Exclusion Criteria:

* Thick hair that makes good measurements difficult/impossible
* obvious malformations or syndromes
* Complications in relation to caesarean section
* Depression after birth (APGAR < 8 after 1 minute)

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term infants born by elective caesarean section at Rigshospitalet, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | 10 minutes
  The sensors of both instruments will be placed on each side of the head. They will be held by hand by self-adhesive tape as appropriate.

SECONDARY OUTCOMES:
Reproducibility | 10 minutes
  The sensor will be placed 6 times alternating on each frontoparietal region and held by hand, obtaining 30 seconds of signal for each placement. The placements will be in the same region but not in exactly the same spot. This will be done for both devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Gorm Greisen, Copenhagen, Copenhagen, Denmark